CLINICAL TRIAL: NCT00487786
Title: A Phase 1 Study Evaluating A Second Generation Antisense Oligonucleotide (OGX 427) That Inhibits Heat Shock Protein 27 (Hsp27
Brief Title: Safety Study of an Antisense Product in Prostate, Ovarian, NSCL, Breast or Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OGX-427-01
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2014-04

CONDITIONS: Neoplasms
Keywords: Antisense; Heat Shock Protein
MeSH Terms: conditions — Neoplasms | interventions — apatorsen; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Each patient receives OGX-427
  Interventions: Drug: OGX-427; Drug: Docetaxel

INTERVENTIONS:
Drug: OGX-427 — OGX-427 injection at 200mg, 400mg, 600mg, 800mg or 1000mg once a week until withdrawn
Drug: Docetaxel — injection - 75 mg/M2 IV on Day 1 every 21 days for cohorts 6 & 7 only, together with appropriate dose of OGX-427 until withdrawn from study
  Other Names: Taxotere

SUMMARY:
This study is for patients with cancer who have failed potentially curative treatments or for whose disease a curative treatment does not exist.

OGX-427 is an antisense product that inhibits expression of one of the heat shock proteins. Decreasing this heat shock protein (Hsp27) should result in down regulation of pathways implicated in cancer progression and development of resistance to treatment.

DETAILED DESCRIPTION:
This study is for patients with breast, prostate, ovarian, non-small cell lung (NSCL) or bladder cancer who have failed potentially curative treatments or for whose disease a curative treatment does not exist.

OGX-427 is a second-generation ASO that inhibits expression of Hsp27. Hsp27 is one of the heat shock proteins. Hsp27 increases with cell stress, including cytotoxic chemotherapy, radiation therapy and hormone therapy and has been shown to inhibit cell death. Thus, decreasing Hsp27 as a cancer therapy is attractive as a therapy as it should result in down regulation of pathways implicated in cancer progression and development of resistance to treatment.

A number of in vitro and in vivo pharmacological studies have demonstrated that OGX-427 has single-agent activity in reducing Hsp27, inhibiting cell growth and inducing cell death in several human cancer cell lines. OGX-427 has also demonstrated chemosensitizing activity in studies using cell lines and animal models in combination with several cytotoxic drugs, including docetaxel.

Docetaxel (Taxotere®) has anticancer activity in breast, prostate, ovarian, non-small cell lung and bladder cancer. Docetaxel has been approved by Health Canada and the Food and Drug Administration for the treatment of patients with breast, prostate, ovarian and non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years at time of consent.
* Histologically or cytologically confirmed diagnosis of one of the following: adenocarcinoma of the breast, ovary, or prostate, any NSCLC or bladder cancer.
* Must have metastatic disease. Prostate cancer patients must be hormone refractory.
* Must have failed therapies that are potentially curative; failed/refused standard therapy known to prolong survival or progression-free survival; or failed/refused therapy, that in the view of the investigator, would be beneficial in improvement of symptoms
* Patients enrolled into Cohorts 6 and 7 (OGX 427 in combination with docetaxel) must have disease that has a possibility of responding to docetaxel.
* A minimum of 28 days must have elapsed between any major surgery, the last dose of chemotherapy, radiotherapy (except limited fields-see #7 below), radioisotope, immunotherapy or experimental agent and enrollment onto the study. Note: Patients on hormone or estrogen therapy and steroids for treatment of their disease may remain on therapy.
* A minimum of 7 days must have elapsed between a single fraction of ≤ 800 cGy to a limited field or conventional radiotherapy to a limited non marrow-bearing field such as an extremity or orbit and enrollment onto the study.
* Recovery from all toxicities of prior therapy including chemotherapy, radiation therapy, immunotherapy and experimental agents to ≤ grade 2 by NCI CTCAE, version 3.0.
* If not treated with bilateral orchiectomy, patients with HRPC must be willing to continue luteinizing hormone releasing hormone (LHRH) analogues throughout the study.
* If taking opioid medication, patient must be willing to continue on the same opioid medication that they are on at enrollment through the PK/ECG evaluations during Cycle 1.
* Karnofsky score of ≥60%.
* Various laboratory requirements.
* Must be willing to use effective contraception during and for 3 months following treatment if of child bearing potential.
* Must be willing to undergo pharmacokinetic blood draws and frequent ECG monitoring on Days 1 and 2 of Cycle 1.
* Must provide written, informed consent.

Exclusion Criteria

* More than three cytotoxic chemotherapy regimens.
* Current treatment with any anticancer agent including but not limited to trastuzumab, aromatase inhibitors, or tamoxifen. Steroids, bisphosphonates and female hormone replacement therapy are allowed.
* Documented central nervous system (CNS) metastasis or carcinomatous meningitis.
* For patients in Cohorts 6 and 7, prior history of a serious allergic reaction to docetaxel; any chemotherapy containing Cremophor EL (used in drugs such as cyclosporine, etoposide, teniposide); or polysorbate 80 (the diluent for docetaxel).
* Current pregnancy or lactation.
* Current second malignancy except for non melanoma skin cancers, superficial bladder cancer, early cervical cancer or early prostate cancer not requiring treatment.
* Uncontrolled and/or serious medical conditions such as, but not limited to, active infection, symptomatic congestive heart failure, unstable angina, significant cardiac arrhythmia, significant neurological dysfunction, history of myocardial infarction or stroke within the 3 months prior to enrollment or any other condition which the Investigator feels would preclude protocol therapy.
* Concomitant participation in another clinical trial of an experimental drug, vaccine or device.
* Prior high dose chemotherapy requiring stem cell rescue.
* Atrial fibrillation, left bundle branch block, or obligatory use of a cardiac pacemaker.
* Currently on a drug known to increase the QTc duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
• To determine the maximum tolerated dose (MTD) of OGX-427 when administered as a single agent, up to a 1000 mg dose level. | approximately 2 years
• To further evaluate the safety profile at one dose level below the MTD derived for OGX-427 administered as a single agent and at the MTD level when OGX 427 is administered in combination with a taxane chemotherapy (docetaxel). | approximately 2 years

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of OGX-427 when used as a single agent and when used in combination with a taxane. | approximately 2 years
To determine whether OGX-427 alone or when co-administered with a taxane alters ECG intervals and morphology. | approximately 2 years
To document objective responses and disease stabilization when OGX-427 is administered either alone or in combination with a taxane. | approximately 2 years
To assess for a biologically effective dose(s) of OGX-427 that inhibits Hsp27 and other related protein levels in patient's serum. | approximately 2 years
To assess for a biologically effective dose(s) of OGX-427 when used as a single agent that reduces serum PSA levels in patients with HRPC. | approximately 2 years
To estimate a biological dose with an acceptable toxicity profile for further evaluation in Phase 2 studies | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kim Chi, M.D., Principal Investigator — University of British Columbia
Locations (3):
- Seattle Cancer Care Alliance, Seattle, Washington, United States
- Canada (2):
  - BC Cancer Agency, Vancouver, British Columbia
  - Juravinski Cancer Center, Hamilton, Ontario

REFERENCES:
- [Derived] Chi KN, Yu EY, Jacobs C, Bazov J, Kollmannsberger C, Higano CS, Mukherjee SD, Gleave ME, Stewart PS, Hotte SJ. A phase I dose-escalation study of apatorsen (OGX-427), an antisense inhibitor targeting heat shock protein 27 (Hsp27), in patients with castration-resistant prostate cancer and other advanced cancers. Ann Oncol. 2016 Jun;27(6):1116-1122. doi: 10.1093/annonc/mdw068. Epub 2016 Feb 18. PMID 27022067